CLINICAL TRIAL: NCT02720354
Title: A Phase I Study of a Novel Tracer for Positron Emission Tomography "PET" Myocardial Perfusion Imaging "MPI"
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Synektik S.A. (Industry)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SK-DMDPA-001
Record Dates: First submitted 2016-03-15; First posted 2016-03-25 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2016-11

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A single Intravenous bolus injection (Experimental): A single Intravenous bolus injection of 11C[DMDPA]
  Interventions: Other: [11C]-DMDPA

INTERVENTIONS:
Other: [11C]-DMDPA

SUMMARY:
[11C]-dimethyl-diphenyl ammonium ([11C]-DMDPA) - A Phase I, Open-label, Safety and Tolerability, Radiation Dosimetry, Biodistribution, First-in-Human Study of a Novel 11C-labeled Tracer for Positron Emission Tomography Myocardial Perfusion Imaging

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) between 18.0 and 30.0 kg/m2
* good health
* written informed consent

Exclusion Criteria:

* smokers
* subject receiving medication
* a blood transfusion in the 4 weeks prior to screening
* positive alcohol blood test
* Subjects who suffer from claustrophobia
* Subjects who have had a clinically significant illness
* Subjects exposed to radiation within 12 months prior to screening

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Measurement of absorbed radiation dose for all target organs in megabecquerel (the activity of a quantity of radioactive material in which one nucleus decays per second). | within 80 minutes